CLINICAL TRIAL: NCT00586365
Title: Effectiveness of Naproxen for the Prevention of Heterotopic Ossification After Complex Elbow Trauma: a Prospective Randomized Trial
Brief Title: Naproxen for the Prevention of HO After Complex Elbow Trauma
Acronym: Naproxen
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Too difficult to satisfy all the inclusion criteria.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Director of Research, Hand Service, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006-P-001670
Record Dates: First submitted 2007-12-14; First posted 2008-01-04 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Heterotopic Ossification
Keywords: complex elbow trauma; prevention; complication; naproxen; NSAIDS
MeSH Terms: conditions — Ossification, Heterotopic | interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Will receive 500 mg Naproxen twice a day for two weeks
  Interventions: Drug: Naproxen
- 2 (No Intervention): Will not receive naproxen

INTERVENTIONS:
Drug: Naproxen — 500 mg Naproxen twice a day for two weeks
  Arms: 1

SUMMARY:
Complex elbow fractures can lead to formation of new bone (called Heterotopic ossification). This new bone is unwanted and it can restrict motion. This research study is being done to learn more about the effect of the drug naproxen, on unwanted formation of new bone around the elbow as it heals after a fracture. Naproxen belongs to a class of drugs called NSAIDs which stands for non-steroidal anti-inflammatory drugs.

Several research studies suggest that NSAIDs such as Naproxen can prevent the unwanted formation of new bone around the hip. The effect of NSAIDS on the formation of bone around the elbow has not been studied as well as it has been studied for their effect on the hip.

The drug, Naproxen is approved by the US food and drug administration (FDA) for sale but ot specifically for the treatment of heterotopic ossification.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 years or greater
2. Operative treatment of one of the following injuries

   * An elbow dislocation with or without associated fractures
   * An olecranon fracture-dislocation, but not simple olecranon fractures
   * A distal humerus fracture

Exclusion Criteria:

1. An existing diagnosis of one of the following conditions

   * Injury to the central nervous system, thorax, or abdomen precluding the immediate use of non-steroidal anti-inflammatory medications
   * Fracture of any long bone since non-steroidal anti-inflammatory medications may increase the risk of nonunion
   * History of gastritis, peptic ulcer disease, or upper gastrointestinal bleeding
   * Impaired renal function (creatinine > 2.0), hypovolemia, heart failure, high blood pressure ( > 160/90), fluid retention, asthma, liver dysfunction (bilirubin > 2.0), or a coagulation disorder
   * Allergy to non-steroidal anti-inflammatory medications
   * Asthma, nasal polyps, urticaria, and hypotension associated with the use of NSAIDs
   * Considerable dehydration
2. Pregnant or breast-feeding women
3. Concomitant use of one of the following drugs:

   * Aspirin
   * Other naproxen products (ec-naprosyn, anaprox, anaprox ds, naprosyn suspension, aleve)
   * Methotrexate
   * Diuretics (thiazides / furosemide)
   * ACE-inhibitors (captopril, enalapril, ramipril etc.)
   * Beta-blockers (propanolol etc.)
   * Probenecid (for gout or hyperuricemia)
   * H2-blockers, sucralfate and intensive antacid therapy
   * Lithium
   * Anticoagulants / Warfarin (coumadin, waran, jantoven etc.)
   * Sulfonamides
   * Anticonvulsant medication (peganone, mesantoin, cerebyx, dilantin, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
There is no difference in ulnohumeral flexion | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD PhD, Study Director — Mass General
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Viola RW, Hastings H 2nd. Treatment of ectopic ossification about the elbow. Clin Orthop Relat Res. 2000 Jan;(370):65-86. doi: 10.1097/00003086-200001000-00008. PMID 10660703